CLINICAL TRIAL: NCT02850926
Title: The Effectiveness of Soccer Headgear to Reduce Concussion in Adolescents
Brief Title: Effect of Soccer Head Gear to Reduce Concussions
Acronym: Socheadgear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Operating Committee on Standards for Athletic Equipment (NOCSAE) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MSN186953
Record Dates: First submitted 2016-07-25; First posted 2016-08-01 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Brain Concussion
Keywords: Concussion; Soccer; Adolescent
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Soccer head gear (Experimental): Subjects who are wearing soccer head gear during the practices and games during the soccer season.
  Interventions: Other: Soccer head gear
- Control (No Intervention): Subjects who are not wearing soccer head gear during the practices and games during the soccer season.

INTERVENTIONS:
Other: Soccer head gear — Each head gear model consists of lightweight materials with a cross strap design that is fully adjustable or a single elastic headband. All models meet or exceed the American Society for Testing and Materials (ASTM) testing standards for soccer headgear and are approved by the National Federation of High Schools and The Fédération Internationale de Football Association (FIFA) for use by interscholastic soccer players. Players will be allowed to choose the brand of head gear to use and wear it for each practice and game during the soccer season.
  Arms: Soccer head gear

SUMMARY:
This study will determine if protective soccer headgear reduces the incidence or severity of Sport Related Concussion injuries (SRCs) in US adolescent (high school) soccer players. Half the subjects will practice and play during their soccer season with soccer head gear specifically marketed to reduce the incidence of SRCs while the other half of the subjects will practice and play without the head gear.

DETAILED DESCRIPTION:
High school soccer is a very popular sport, with over one million male and female participants nationwide each year. Approximately 109,000 Sport Related Concussion SRCs were sustained by U.S. high school soccer players last year.

Despite the high incidence of SRCs in this population, little is known about the type of protective head gear that is being marketed to players and coaches to prevent SRCs. There are conflicting lab studies that show players may or may not be protected from sustaining a SRC while wearing head gear. However, there have been no large, prospective, randomized trials to examine the effect of soccer headgear on the incidence and severity of SRC in high school soccer players.

Approximately 3,000 high school soccer players (male and female, age 14-18, grades 9 - 12) from 88 United States high schools (44 per year) will be enrolled as subjects. All subjects will be asked to complete a short baseline survey regarding their previous history of SRCs. Schools will be randomly assigned to be in the head gear (intervention) group or no head gear (control) group. Subjects in schools assigned to the intervention group (n = 1500, 44 schools) will be asked to wear the protective soccer head gear provided by the study team for all practices and games throughout their high school soccer season. Subjects in the control group schools (n = 1500, 44 schools) will be allowed to practice and compete as they normally would (without head gear). Licensed athletic trainers (ATs) employed at each participating school will electronically record and report the characteristics of all SRCs that are sustained by the subjects as well as their athletic exposures to the study team.

At the conclusion of the data collection, the rate of SRCs will be estimated using Kaplan and Meier survival analysis and compared between the intervention and control group using a log-rank test. Cox Proportional Hazards modeling will be utilized to examine the relationship between SRCs and the independent variables (age, sex, competition level and previous SRC history). Wilcoxon Rank Sum tests will be used to determine if there was a significant difference in the injury severity between the intervention and control subjects. All analyses will control for school cluster effect and will be performed at the threshold of α = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* be a member on one (freshman, junior varsity or varsity) of the schools interscholastic soccer teams
* be in grades 9 to 12,
* be able to fully participate (no disabling injuries) in team activities on the day of pre-season team practices
* athlete and parent (when appropriate) sign the mandated University of Wisconsin Research Informed Assent/Consent and HIPAA Research Forms.

Exclusion Criteria:

* are not a member of the schools interscholastic soccer (freshman, junior varsity or varsity) teams,
* are not in grades 9 to 12,
* the athlete or parent (when appropriate) does not sign the mandated University of Wisconsin Research Informed Assent/Consent and HIPAA Research Forms.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3050 (Actual)
Dates: Start 2016-08; Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
The number Sport Related Concussion injuries | 2 years
  To determine if the number of SRC injuries in soccer players wearing HG is lower than soccer players who did not wear head gear (NoHG).

SECONDARY OUTCOMES:
Number of days of soccer participation lost due to Sport Related Concussion injuries | 2 years
  To determine if the average number of days of soccer participation lost post Sport Related Concussion injury is different between soccer players in the HG group compared to players in the NoHG group.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A McGuine, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] McGuine T, Post E, Pfaller AY, Hetzel S, Schwarz A, Brooks MA, Kliethermes SA. Does soccer headgear reduce the incidence of sport-related concussion? A cluster, randomised controlled trial of adolescent athletes. Br J Sports Med. 2020 Apr;54(7):408-413. doi: 10.1136/bjsports-2018-100238. Epub 2019 May 14. PMID 31088784